CLINICAL TRIAL: NCT05631301
Title: Move&Connect: A Holistic Interdisciplinary Program of Care for Youth Experiencing Persistent Symptoms Post-concussion and Their Caregivers
Brief Title: Move&Connect: A Program for Youth With Concussion and Their Caregivers.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Shannon Scratch, Clinical Neuropsychologist, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-0513
Record Dates: First submitted 2022-10-28; First posted 2022-11-30 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Post-Concussion Syndrome
Keywords: Concussion; Rehabilitation; Exercise; Education
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Concussion; Motor Activity | interventions — Organizational Objectives

STUDY DESIGN:
Intervention Model Description: The M&C-Youth & M&C-Caregiver intervention will both run for six weeks in one of three groups (Two treatments: direct, virtual; One control: waitlist). The treatment sessions run once a week and last approximately one hour. Individuals initially enrolled in the waitlist control arm will be subsequently be invited to participate in the intervention arm of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Move&Connect-Youth (Experimental): * Sessions run weekly at the Bloorview Research Institute by a registered physiotherapist and occupational therapist for one hour. Participants will provide electronic consent and complete the pre-intervention measures one week before the intervention begins. Data collection will also occur on week 8 (post intervention) and at 3-month follow-up.
  * Weekly sessions will include an active rehabilitation component including exercises focused on cardiovascular fitness, balance, co-ordination and strength.
  * Weekly sessions will also include an educational component through focused discussions on topics including headache management, stress coping skills, fatigue management, advocacy skills, and goal setting.
  * Data collection sessions will include a series of questionnaires and surveys to acquire consent, demographic information, and assess pre-post changes in concussion symptoms, self-efficacy, quality of life, mental health and social support.
  Interventions: Other: Exercise Circuits; Behavioral: Goal Setting; Behavioral: Psychoeducation-Youth
- Move&Connect-Youth-Virtual (Experimental): * Sessions run weekly via Zoom videoconferencing by a registered physiotherapist and occupational therapist for one hour. Participants will provide electronic consent and complete the pre-intervention measures one week before the intervention begins. Data collection will also occur on week 8 (post intervention) and at 3-month follow-up.
  * Weekly sessions taking place over Zoom will include an active rehabilitation component including exercises focused on cardiovascular fitness, balance, co-ordination and strength.
  * Weekly sessions will also include an educational component through focused discussions on topics including headache management, stress coping skills, mood coping skills, fatigue management, advocacy skills, and goal setting.
  * Data collection sessions will include a series of questionnaires and surveys to acquire consent, demographic information, and assess pre-post changes in concussion symptoms, self-efficacy, quality of life, mental health and social support.
  Interventions: Other: Exercise Circuits; Behavioral: Goal Setting; Behavioral: Psychoeducation-Youth
- Move&Connect-Youth Waitlist control (Other): The control group will be recruited from the waitlist for the Persistent Concussion Clinic and the Early Care Concussion Clinic at Holland Bloorview, in addition to partnered community medical offices and organizations.
  For the control group, the research assistant will schedule the participants first session to obtain consent and provide youth/caregivers with week 1 questionnaires. At this time, the participants will be able to ask any questions related to the study. After eight weeks the control group will be asked to complete the post measures in order to mimic the length of the intervention. The control group will then be given the opportunity to enroll in one of the intervention arms of the Move&Connect study. They will then follow the same approved procedures for the intervention treatment group. Youth and their caregivers will be able to participate as waitlist controls without completing the intervention, if they choose.
  Interventions: Other: Waitlist Control Surveys
- Move&Connect-Caregiver (Experimental): * The treatment sessions run once a week at the Bloorview Research Institute and last approximately one hour. Participants will provide electronic consent and complete the pre-intervention measures one week before the intervention begins. Data collection will also occur on week 8 (post intervention) and at 3-month follow-up.
  * Caregivers will participate in a group-based psychoeducational support group with sessions consisting of focused discussions on topics including: the ripple effect, school advocacy, child well-being, family functioning, parenting, and stress & daily challenges. The sessions will be run by a clinical neuropsychologist and social worker.
  * Data collection sessions will include a series of questionnaires and surveys to acquire consent, demographic information, and assess pre-post changes in their youth's concussion symptoms, and mental health, as well as parental self-efficacy, quality of life, mental health and social support.
  Interventions: Behavioral: Psychoeducation-Caregiver
- Move&Connect-Caregiver-Virtual (Experimental): * The treatment sessions run once a week using Zoom videoconferencing and last approximately one hour. Participants will provide electronic consent and complete the pre-intervention measures one week before the intervention begins. Data collection will also occur on week 8 (post intervention) and at 3-month follow-up.
  * Caregivers will participate in a group-based psychoeducational support group with sessions consisting of focused discussions on topics including: the ripple effect, school advocacy, child well-being, family functioning, parenting, and stress & daily challenges. The sessions will be run by a clinical neuropsychologist and social worker.
  * Data collection sessions will include a series of questionnaires and surveys to acquire consent, demographic information, and assess pre-post changes in their youth's concussion symptoms, and mental health, as well as parental self-efficacy, quality of life, mental health and social support.
  Interventions: Behavioral: Psychoeducation-Caregiver
- Move&Connect-Caregiver Waitlist control (Other): The control group will be recruited from the waitlist for the Persistent Concussion Clinic and the Early Care Concussion Clinic at Holland Bloorview, in addition to partnered community medical offices and organizations.
  For the control group, the research assistant will schedule the participants first session to obtain consent and provide youth/caregivers with week 1 questionnaires. At this time, the participants will be able to ask any questions related to the study. After eight weeks the control group will be asked to complete the post measures in order to mimic the length of the intervention. The control group will then be given the opportunity to enroll in one of the intervention arms of the Move&Connect study. They will then follow the same approved procedures for the intervention treatment group. Youth and their caregivers will be able to participate as waitlist controls without completing the intervention, if they choose.
  Interventions: Other: Waitlist Control Surveys

INTERVENTIONS:
Other: Exercise Circuits — Weekly exercise circuits with a focus on strength, balance, cardiovascular fitness, and coordination
  Arms: Move&Connect-Youth; Move&Connect-Youth-Virtual
Behavioral: Goal Setting — Goal setting focused on the management of persistent post concussion symptoms, exercise, and engagement in daily activities
  Arms: Move&Connect-Youth; Move&Connect-Youth-Virtual
Behavioral: Psychoeducation-Youth — Targeted educational sessions with a focus on the physical, cognitive, and psychological implications of persistent post-concussion symptoms.
  Arms: Move&Connect-Youth; Move&Connect-Youth-Virtual
Behavioral: Psychoeducation-Caregiver — Psychoeducational sessions focused on social support, in addition to addressing the implications of caring for youth experiencing persistent post concussion symptoms
  Arms: Move&Connect-Caregiver; Move&Connect-Caregiver-Virtual
Other: Waitlist Control Surveys — Surveys completed in week 1, and 8 for a subset of participants who are not involved in the study intervention to mirror study timeline and serve as control data for outcome measures assessed during experimental intervention
  Arms: Move&Connect-Caregiver Waitlist control; Move&Connect-Youth Waitlist control

SUMMARY:
Move&Connect is an interdisciplinary group-based program co-designed with youth and caregivers that provides skills training, mental health support, and psychoeducation to caregivers and combines these tenets with active rehabilitation for youth with concussion.

DETAILED DESCRIPTION:
The overall purpose of this project is to pilot the Move&Connect intervention to examine intervention effects of both Move&Connect youth (M&C-Y) and caregiver (M&C-C) arms in comparison to waitlist control when conducted either virtually or in-person.

M&C-Y is a group-based exercise (active rehabilitation) program designed for youth with persistent post-concussion symptoms (PPCS) to exercise, learn new skills to manage concussion symptoms in daily life, and meet others with similar experiences. Program elements include: Goal setting, icebreakers, a circuit exercise program, and psychoeducation about concussion and symptoms. M&C-Y will be delivered/supervised by an Occupational Therapist and Physiotherapist with experience working with youth with concussion.

M&C-C is a group-based psychoeducational support group designed for caregivers who have a child experiencing PPCS. It is designed to provide education centered around advocacy skills, familial and child well-being, and parenting support. M&C-C will be delivered by a Clinical Neuropsychologist and Social Worker with experience working with youth with concussion.

The M&C-Y & M&C-C intervention will both run for six weeks in one of three conditions ((1) direct treatment; (2) virtual treatment; (3) waitlist control). The treatment sessions run once a week and last approximately one hour. Participants will provide electronic consent and complete the pre-intervention (baseline/week 1) measures one week before the intervention begins. Data collection will also occur post-intervention (week 8) and at 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria Youth:

* Between the ages of 8-21 years old with capacity to provide consent/assent.
* Diagnosed with a concussion by a physician or nurse practitioner and are experiencing concussion symptoms for ≥ 4 weeks post concussion.
* Willing to engage in weekly sessions
* Have access to reliable internet connection.

Inclusion Criteria Caregivers:

* Caregiver to youth experiencing PPCS
* Fluent in English
* Have the capacity to consent
* Have access to a reliable internet connection.

Exclusion Criteria Youth:

* Unable to read and speak English
* Unable to provide informed consent.
* Diagnosed with autism spectrum disorder (ASD), a physical disability (requiring a-mobility device) and and/or intellectual disabilities.
* Diagnosed with a functional neurological disorder (e.g. conversion disorder, somatization, personality disorder) or an acute psychiatric condition (e.g. schizophrenia, suicidality, or a recent hospital admission for another psychiatric condition).

Exclusion Criteria Caregivers:

• Diagnosed with an acute psychiatric condition that resulted in a recent hospital admission (e.g. schizophrenia, suicidality, etc.).

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Canadian Occupational Performance Measure at 8 weeks and 3-month follow up | Baseline, 8 weeks, 3-month follow-up
  An evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living (satisfaction in self-care, productivity and leisure). It assists therapists in using a client-centred approach to service delivery by indicating the family's priorities.
Change from baseline Health and Behavior Inventory at 8-weeks and 3-month follow up | Baseline, 8 Weeks, 3-month follow-up
  A 20-item self-report form that focuses on concussion symptoms in the cognitive, emotional, and somatic domains. Questions are scored on a scale from 0-3 with higher scores indicating higher symptom frequency.
Change from baseline Family Assessment Device-General Functioning at 8-weeks and 3-month follow up | Baseline, 8 weeks, 3 month follow-up
  A 12-item measure of family functioning. Each item is a statement about a family and participants rate how well it describes their own family. Each item is scored based on the level of agreement with each statement with four options from strongly agree, to strongly disagree
Change from baseline Patient-Reported Outcomes Measurement Information System Bank v1.0- Depression at 8-weeks and 3-month follow up | Baseline, 8 weeks, 3-month follow-up
  A 28-item self-report form that focuses on negative mood, social cognition and decreased positive affect and engagement. Each item is scored on a scale from 1-5 with higher scores indicating increased frequency of depressive symptoms
Change from baseline Patient-Reported Outcomes Measurement Information System Bank v1.0- Anxiety at 8-weeks and 3-month follow up | Baseline, 8 weeks, 3-month follow-up
  A 29-item self-report form that focuses on feelings of fear, anxiousness, hyperarousal, and somatic symptoms related to arousal. Each item is scored on a scale from 1-5 with higher scores indicating increased frequency of symptoms of anxiety

SECONDARY OUTCOMES:
Semi-Structured Exit Interview | Week 8
  To assess perceived changes in persistent concussion symptoms, education, and social support a participant may/may not have experienced during the intervention and to gather feedback on the structure and delivery of the intervention
Change from baseline Brief Illness Perception Questionnaire at 8-weeks and 3-month follow up | baseline, week 8, 3-month follow-up
  An 8-item questionnaire to assess cognitive and emotional representations of illness.
  Each item represents one domain of illness perception and each item is scored on a scale from 1-10. Items 3,4, and 7 are reverse scored and all scores are added together with a higher score indicating a more threatening view of illness
Change from baseline Patient-Reported Outcomes Measurement Information System Pediatric Bank v2.0- Depression at 8-weeks and 3-month follow up | baseline, week 8, 3-month follow-up
  A 14-item self-report form that focuses on negative mood, social cognition and decreased positive affect and engagement. Each item is scored on a scale from 1-5 with higher scores indicating increased frequency of depressive symptoms
Change from baseline Patient-Reported Outcomes Measurement Information System Pediatric Bank v2.0- Anxiety at 8-weeks and 3-month follow up | baseline, week 8, 3-month follow-up
  A 15-item self-report form that focuses on feelings of fear, anxiousness, hyperarousal, and somatic symptoms related to arousal. Each item is scored on a scale from 1-5 with higher scores indicating increased frequency of symptoms of anxiety
Change from baseline Patient-Reported Outcomes Measurement Information System Pediatric Bank v2.0 Fatigue Short form 10a at 8-weeks and 3-month follow up | baseline, week 8, 3-month follow-up
  Assesses a range of symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion. Each item is scored on a scale from 1-5 with higher scores indicating increased frequency of symptoms of fatigue
Change from baseline Healthy Lifestyle and Behaviours Checklist at 8-weeks and 3-month follow up | baseline, week 8, 3-month follow-up
  A self-report questionnaire of an individual's physical activity, and sleep behaviors.
Change from baseline Progressive Activities of Controlled Exertion- Self Efficacy at 8-weeks and 3-month follow up | baseline, week 8, 3-month follow-up
  A 17-item measure that assesses children's perceptions of self-efficacy for an active approach toward pediatric concussion recovery. Each item is scored on a scale of 1-10 with higher scores indicating greater perceived self efficacy.
Change from baseline University of California, Los Angeles Loneliness Scale at 8-weeks and 3-month follow up | baseline, week 8, 3-month follow-up
  A 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. each item is scored on a scale of 1 (never) to 4 (often). Items 1, 5, 6, 9, 10, 15, 16, 19, 20 are all reverse scored. Higher total scores indicate elevated feelings loneliness and likelihood of interpersonal problems.
Change from baseline Pediatric Quality of Life Index: Generic Core Scales at 8-weeks and 3-month follow up | baseline, week 8, 3-month follow-up
  a 23-item measure that assesses the core dimensions of health as delineated by the World Health Organization including Physical Functioning, Emotional Functioning, Social Functioning and School Functioning. Each item is scored from 0 (never) to 4 (almost always) with higher scores representing worse outcomes in each domain.
Change from baseline Patient-Reported Outcomes Measurement Information System Parent Proxy Bank v2.0-Depressive Symptoms short form 6a at 8-weeks and 3-month follow up | baseline, week 8, 3-month follow-up
  A 6 item parent proxy-report that focuses on negative mood, social cognition and decreased positive affect and engagement in their child. Each item is scored on a scale from 1-5 with higher scores indicating increased frequency of depressive symptoms reported in their child
Change from baseline Patient-Reported Outcomes Measurement Information System Parent Proxy Bank v2.0 - Anxiety short form 8a at 8-weeks and 3-month follow up. | baseline, week 8, 3-month follow-up
  A 8 item parent proxy-report form that focuses on feelings of fear, anxiousness, hyperarousal, and somatic symptoms related to arousal in their child. Each item is scored on a scale from 1-5 with higher scores indicating increased frequency of symptoms of anxiety in their child

OTHER OUTCOMES:
Satisfaction Survey | Week 8
  To collect general feedback related to the structure and delivery of the Move&Connect intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Scratch, PhD, C Psych, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Andrea Hickling, MScOT, OT Reg. (Ont.), Study Director — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, East York, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No